CLINICAL TRIAL: NCT07120061
Title: Test-retest Reliability of the Maintenance of Wakefulness Test in Participants With Hypersomnolence
Acronym: REWIND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Société Française de Recherche et Médecine du Sommeil (S.F.R.M.S) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2024/88
Record Dates: First submitted 2025-07-29; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Disorders of Excessive Somnolence
Keywords: Hypersomnolence; Driving risk; Biomarker; Maintenance of Wakefulness; Test-retest reliability
MeSH Terms: conditions — Disorders of Excessive Somnolence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1a (Experimental): Patient with obstructive sleep apnea (OSA) before/without treatment for OSA
  Interventions: Diagnostic Test: First MWT; Diagnostic Test: second MWT; Device: actimetry
- 1b (Experimental): Patient with obstructive sleep apnea (OSA) treated for OSA
  Interventions: Diagnostic Test: First MWT; Diagnostic Test: second MWT; Device: actimetry
- 2 (Experimental): Participants with type 1 narcolepsy
  Interventions: Diagnostic Test: First MWT; Diagnostic Test: second MWT; Device: actimetry
- 3 (Active Comparator): Healthy volunteers
  Interventions: Diagnostic Test: First MWT; Diagnostic Test: second MWT; Device: actimetry

INTERVENTIONS:
Diagnostic Test: First MWT — MWT during the first visit of the protocol
Diagnostic Test: second MWT — MWT during the second visit of the protocol
Device: actimetry — In order to monitor compliance with the guidelines prior to each MWT, namely good sleep hygiene in the 14 days preceding the MWT, and in accordance with the recommendations of the AASM, an actimeter will be worn by the participant.

SUMMARY:
This study will provide the first measurement of the test-retest reliability of the Maintenance of Wakefulness Test (MWT) with a prospective multicenter design. A high level of reliability will reinforce the place of the MWT as an essential tool to respond to the medical and legal worldwide issue of the driving risk related to hypersomnolence. This would legitimize its place as a medico-legal examination in France and promote its diffusion in other countries. A low level of reliability will call into question the place of the MWT in the management of participants with hypersomnolence. Bordeaux University Hospital is the sponsor of this research. This research will be conducted with the support of Société Française de Recherche en Médecine du Sommeil.

DETAILED DESCRIPTION:
Hypersomnolence is a frequent and disabling symptom that has an impact on an individual's daytime functioning and particularly on driving, increasing the risk of traffic accidents related to sleepiness. Objective markers for assessing hypersomnolence are particularly important to overcome reporting bias since it is listed as a factor of temporary medical incompatibility to obtain or maintain a driving license in several countries, including France. According to the American Academy of Sleep Medicine (AASM), the MWT is the most relevant test for medico-legal assessments of fitness to drive.

Several experimental and epidemiological studies have shown that mean sleep latency at the MWT is a valid biomarker for assessing driving risk. However, there is currently no data on the test-retest reliability of the MWT from one day to the next. This is all the more important given the implications on the driving ability, and the variability associated with good participant compliance (good sleep hygiene the night before the test, absence of stimulation during the test). This study will use a factorial design to allow for stratified analyses with strong power (50 participants with Obstructive sleep apnea syndrome (OSAS), including 25 before/without treatment and 25 after/under treatment, and 25 participants with narcolepsy type 1 ,(after/under treatment) and 25 healthy volunteers. All participants will undergo an inclusion visit (V0) and two MWT (V1 and V2) separated by less than 28 days. All MWT will be twice blinded analyzed by a single expert to minimize variability of interpretation.

ELIGIBILITY:
Inclusion Criteria :

* Being affiliated or beneficiaries of a social security system.
* Having been informed of the study and having given their free and informed consent, written and signed consent to participate to the study

Plus one of the following inclusion criteria:

* Participant with a suspicion of OSAS without any previous diagnosis or treatment and with Epworth Sleepiness Scale ≥ 11.
* Participant with effective and stable treatment for OSAS (defined by apnea-hypopnea index ≥ 15 per hour) since at least 15 days and intended to be explored by a MWT.
* Participant with effective and stable treatment for narcolepsy type 1 as defined by the ICSD-3 (cataplexy or lack of orexine) since at least 15 days and intended to be explored by a MWT.
* Healthy volunteers with Epworth Sleepiness Scale < 11.

Exclusion Criteria:

* Comorbid sleep disorders associated with excessive daytime sleepiness (e.g., OSAS and narcolepsy)
* Severe conditions endangering life in the short term
* Participant with cardiovascular, neurological, psychiatric, respiratory, infectious, endocrine, or systematic pathology, which is not stabilized and may require hospitalization or a modification of therapy during the duration of the study
* Introduction or change in dosage of a psychotropic medication in the previous year which may modify the level of arousal in the previous year and modify the MWT results
* Shift or night workers
* Pregnant or breastfeeding woman
* Participants under curatorship or guardianship

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Mean sleep latency of the MWT | v2 (up to 90 days after V0)
  Sleep latency value in the wakefulness maintenance test.

SECONDARY OUTCOMES:
Bordeaux Sleepiness Scale | at Baseline (day 0), v1 (up to 88 days after day 0) and v2 (up to 90 days after day 0)
  Self-reported traffic accidents or near-misses related to sleepiness and sleepiness at the wheel.
  4-items questionnaire. Total score of 8 points. If the score is 3 or higher, the prediction of the risk of a sleep-related accident or near miss is defined as positive.
Chronotype | at Baseline (day 0), v1 (up to 88 days after day 0) and v2 (up to 90 days after day 0)
  Self-reported chronotype (reduced Morningness-Eveningness Questionnaire) It consists of 5 questions, each with a scoring system ranging from 1 to 5 points (depending on the answers), giving a total score ranging from 4 to 25.
  The lower the score, the more "evening" the chronotype; the higher the score, the more "morning" the chronotype.
Sleepiness (1) | at Baseline (day 0), v1 (up to 88 days after day 0) and v2 (up to 90 days after day 0)
  Self-reported sleepiness using :
  - the Epworth Sleepiness Scale, 8-items, the total score ranges from 0 (normal sleepiness) to 24 (pathological sleepiness)
Sleepiness (2) | at Baseline (day 0), v1 (up to 88 days after day 0) and v2 (up to 90 days after day 0)
  Self-reported sleepiness using :
  - the Hypersomnia Severity Index, 9-items, the total score ranges from 0 (no hypersomnia) to 36 (Very severe Hypersomnia)
Sleepiness (3) | at Baseline (day 0), v1 (up to 88 days after day 0) and v2 (up to 90 days after day 0)
  Self-reported sleepiness using :
  - the Insomnia Severity Index, 7 items, the total score ranges from 0 (no insomnia) to 28 (Severe insomnia)
Sleepiness (4) | at Baseline (day 0), v1 (up to 88 days after day 0) and v2 (up to 90 days after day 0)
  Self-reported sleepiness using :
  - Functional Outcomes of Sleep Questionnaire, 10 items. The total score ranges from 5 ( Significant alteration) to 20 (no alteration)
Quality of life (1) | at Baseline (day 0), v1 (up to 88 days after day 0) and v2 (up to 90 days after day 0)
  Self reported quality of life with :
  - EQ-5D, total score from 0 (Worst possible health) to 100 ( Best possible health)
Quality of life (2) | at Baseline (day 0), v1 (up to 88 days after day 0) and v2 (up to 90 days after day 0)
  Self reported quality of life with :
  - Fatigue Severity Scale, 9 items, total score from 1 (Absence or low fatigue) to 7( Severe fatigue, with marked repercussions)
Quality of life (3) | at Baseline (day 0), v1 (up to 88 days after day 0) and v2 (up to 90 days after day 0)
  Self reported quality of life with :
  - Toronto Hospital Alertness Test, 10 items, total score from 0 (Impaired alertness (low alert)) to 50 (Good vigilance/sufficient alertness)
Sleep behaviors | at Baseline (day 0), v1 (up to 88 days after day 0) and v2 (up to 90 days after day 0)
  Objective sleep behaviors (sleep duration, sleep regularity, sleep timing, using the 2-weeks actigraphy and sleep diary).
Appropriate disorder (1) | at Baseline (day 0), v1 (up to 88 days after day 0) and v2 (up to 90 days after day 0)
  Self-reported severity scale for appropriate disorder using :
  * The Patient Reported Apnea Questionnaire, 16 items (from 0 to 5), The higher the score, the greater the negative impact of Obstructive Sleep Apnea.
  * The Narcolepsy Severity Scale, 15 items, the higher the score, the more severe the symptoms.
Appropriate disorder (2) | at Baseline (day 0), v1 (up to 88 days after day 0) and v2 (up to 90 days after day 0)
  Self-reported severity scale for appropriate disorder using :
  - The Narcolepsy Severity Scale, 15 items, the higher the score, the more severe the symptoms.
Mental complaints (1) | at Baseline (day 0), v1 (up to 88 days after day 0) and v2 (up to 90 days after day 0)
  Mental complaints using :
  - The Generalized Anxiety Disorder-7, 7 items, total score from 0 (no anxiety) to 21(severe anxiety)
Mental complaints (2) | at Baseline (day 0), v1 (up to 88 days after day 0) and v2 (up to 90 days after day 0)
  Mental complaints using :
  - The Perceived Stress Scale, 10 items, total score from 0 (Low stress) to 40 (High stress)
Mental complaints (3) | at Baseline (day 0), v1 (up to 88 days after day 0) and v2 (up to 90 days after day 0)
  Mental complaints using :
  - The Psychological-Physical-Pain Visual Analogue Scale, 3 items from 0 (no pain) to 100 (maximal pain)
Mental complaints (4) | at Baseline (day 0), v1 (up to 88 days after day 0) and v2 (up to 90 days after day 0)
  Mental complaints using :
  - The Adult Self-Report Scale, 18 items, total score from 0(no symptom) to 72 (very frequent/severe symptoms)
Mental complaints (5) | at Baseline (day 0), v1 (up to 88 days after day 0) and v2 (up to 90 days after day 0)
  Mental complaints using :
  - The Participant Health Questionnaire-9, 9 items, total score from 0(no depression) to 27 (severe depression)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Arthur MICOULAUD-FRANCHI, Pr, Principal Investigator — University Hospital, Bordeaux; Julien COELHO, Dr, Study Chair — University Hospital, Bordeaux
Locations (4):
- France (4):
  - CHU de Bordeaux, Bordeaux
  - CHU de Montpellier, Montpellier
  - APHP - Hôtel-Dieu, Paris
  - APHP - la Pitié-Salpêtrière, Paris

IPD SHARING:
Plan to Share IPD: No